CLINICAL TRIAL: NCT05925309
Title: Preventive Effect of Prophylactic Oral Antibiotics Against Cholangitis After Kasai Portoenterostomy in Biliary Atresia: a Randomized Controlled Trial
Brief Title: Preventive Effect of Prophylactic Oral Antibiotics Against Cholangitis After Kasai Portoenterostomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PACK
Record Dates: First submitted 2023-06-14; First posted 2023-06-29 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Biliary Atresia; Cholangitis; Anti-Bacterial Agents
MeSH Terms: conditions — Biliary Atresia; Cholangitis | interventions — Ursodeoxycholic Acid; Methylprednisolone; Fumigant 93; Imipenem; Meropenem; Trimethoprim, Sulfamethoxazole Drug Combination; Cefaclor

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Antibiotics group (Active Comparator): Basic treatment + Prophylactic oral antibiotics
  Interventions: Drug: Basic treatment: sulperazone + ursodeoxycholic acid + compound glycyrrhizin + methylprednisolone + vitamin AD , D , E , K + imipenem or meropenem; Drug: Prophylactic oral antibiotics: compound sulfamethoxazole tablet (SMZ/TMP) + cefaclor
- Non-antibiotics group (Experimental): Basic treatment
  Interventions: Drug: Basic treatment: sulperazone + ursodeoxycholic acid + compound glycyrrhizin + methylprednisolone + vitamin AD , D , E , K + imipenem or meropenem

INTERVENTIONS:
Drug: Basic treatment: sulperazone + ursodeoxycholic acid + compound glycyrrhizin + methylprednisolone + vitamin AD , D , E , K + imipenem or meropenem — Sulperazone 50mg/kg q8h is used intravenously from the first day to the 14th day after KP surgery. Ursodeoxycholic acid 20mg/kg/d p.o, starting from the 5th day after surgery for at least 2 years. Compound glycyrrhizin 20mg/d i.v, 1-4 days after operation, then switch to compound glycyrrhizin tablets 12.5mg b.i.d p.o until 6 months after KP. Methylprednisolone start at 4mg/kg/d i.v on the 8th day after operation, and decrease by 1mg/kg/d every three days. Starting at about the 15th day after operation, methylprednisolone 4mg/kg is given orally every other day, and the dose is gradually reduced at 10-12 weeks. Vitamin AD , D , E , K, are given orally from the 5th day after the KP for at least 2 months. Treatment of cholangitis: sulperazone 50mg/kg q8h i.v., and methylprednisolone could be used. If cholangitis is not controlled, imipenem or meropenem may be used.
Drug: Prophylactic oral antibiotics: compound sulfamethoxazole tablet (SMZ/TMP) + cefaclor — Compound sulfamethoxazole tablet (SMZ/TMP) 25 mg/kg/d p.o. and cefaclor 12.5 mg/kg/d p.o. alternately every 2 weeks, from post-operation day 15 to month 6.
  Arms: Antibiotics group

SUMMARY:
This study is non-inferiority trial design. This study aimed to investigate the effect of prophylactic oral antibiotics on preventing cholangitis in biliary atresia (BA) patients after Kasai portoenterostomy (KP) by comparing the cholangitis rate in BA patients who received prophylactic oral antibiotics and those who did not. The patients were followed up for 2 years after KP.

DETAILED DESCRIPTION:
Biliary atresia (BA) is a devastating inflammatory obstructive neonatal disease affecting intrahepatic and extrahepatic bile ducts. Kasai portoenterostomy (KP) is the mainstay of treatment for BA. Cholangitis is a common complication after KP, with an overall incidence of 22-93%, and an incidence of 30-70% within 6 months after KP. The mechanism of cholangitis may be intestinal bacteria ascending into the intrahepatic biliary system or bacterial colonization, etc. Common causative organisms include Klebsiella, Escherichia coli, Pseudomonas aeruginosa, Enterobacter cloacae, Acinetobacter baumannii, Streptococcus, and Salmonella typhi. There is some controversy about prophylactic antibiotics after KP, and the type, dosage and course of antibiotics in medical institutions around the world vary greatly. After years of improvement, although the postoperative management and short-term prognosis of BA have improved, the overall incidence of cholangitis has not changed much. High-quality evidence for antibiotic prophylaxis after KP remains lacking. It still remains unknown that whether long-term prophylactic oral antibiotics could benefit the patients. Long-term use of antibiotics may not only increase the burden of liver dysfunction in patients, but also lead to antibiotic resistance, intestinal flora disturbance, and increase the risk of allergies and autoimmune diseases. It is of great significance to use evidence-based medicine to find a relatively reasonable cholangitis prevention program.

This study is non-inferiority trial design. This study aimed to investigate the effect of prophylactic oral antibiotics on preventing cholangitis by comparing the cholangitis rate in BA patients who received prophylactic oral antibiotics after KP and those who did not. Patients diagnosed with type III BA and receiving KP at Children's Hospital of Fudan University will be assigned to 2 groups. Both groups received the same basic treatment, then the patients in the antibiotics group received prophylactic oral antibiotics until the 6th month after KP, while the non-antibiotics group no longer used prophylactic antibiotics until cholangitis occurred. The cholangitis rate within 6 months after KP were measured to evaluate the preventive effect of prophylactic oral antibiotics on cholangitis. The patients were followed up for 2 years after KP.

ELIGIBILITY:
Inclusion Criteria:

* Patients whose age of operation is 14-90 d. Sex and race are not restricted;
* Patients who are born with gestational age older than 36 weeks;
* Patients whose body weight before operation > 2 kg;
* Patients diagnosed of type-III BA and underwent KP in Children's Hospital of Fudan University;
* The type-III BA diagnosis is based on cholangiography or operation;
* Patients whose histological features of liver biopsies are reported. HE staining and Masson staining are required, and edema, inflammation, fibrosis, and hyperplasia of intrahepatic bile duct should be reported;
* Patients who are not allergic to postoperative medications;
* Patients who haven't accepted other antibiotic or probiotic therapy.

Exclusion Criteria:

* Patients with cholestasis of non-BA disease;
* Patients who have undergone KP at other institutions;
* Patients whose pathohistological diagnosis is in doubt;
* Patients who undergo liver transplantation immediately after KP;
* Patients with other liver diseases or severe complications (e.g., severe pulmonary hypertension, renal failure, intracranial hemorrhage, etc.) requiring surgical intervention or other medical therapy;
* Patients with severe cardiac, renal, or central nerve system malformations (e.g., tetralogy of Fallot, transposition of the great arteries, cerebral dysplasia, etc.) and have poor prognosis;
* Patients judged by the researchers that they can not comply with the study requirements.

Ages: 14 Days to 90 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 356 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
The occurrence of cholangitis (confirmed or suspected) within 6 months after KP | 6 months after KP
  Definition of cholangitis:
  A. Clinical elements
  1. Fever and/or shivering;
  2. Stool color change;
  3. New/increasing jaundice;
  4. Abdominal discomfort: vomiting, poor, feeding, irritability.
  B. Laboratory and imaging elements
  1. Inflammatory response (WBC and/or CRP and/or PCT);
  2. Increased/increasing transaminases;
  3. Increased/increasing GGT and/or bilirubin;
  4. Bile lakes.
  Suspected cholangitis: one item in A + one item in B. Confirmed cholangitis: two items in A + two items in B or "suspected cholangitis" + positive blood culture.
  The diagnosis of cholangitis requires the exclusion of definite infections of other systems.

SECONDARY OUTCOMES:
The occurrence of cholangitis (confirmed or suspected) within 1 year after KP | 1 year after KP
  The definition of cholangitis is the same as primary outcome.
The occurrence of jaundice clearance within 6 months after KP | 6 months after KP
  Jaundice clearance is defined as total bilirubin (TB) less than 20 μmol/L.
The occurrence of jaundice clearance within 1 year after KP | 1 year after KP
  Jaundice clearance is defined as TB less than 20 μmol/L.
The number of cholangitis recurrence within 6 months after KP | 6 months after KP
  The definition of cholangitis is the same as primary outcome.
The number of cholangitis recurrence within 1 year after KP | 1 year after KP
  The definition of cholangitis is the same as primary outcome.
The patient survive with native liver or not within 2 years after KP | 2 years after KP
The weight gain of the patients from pre-operation to 6 months post KP | From pre-operation to 6 months post KP
  Weight for height (length) Z-score is calculated based on the gender, age, and weight reference standards for children in China. The difference in weight for height (length) Z-score between pre-operation and 6 months post KP is regarded as weight gain.
The weight gain of the patients from pre-operation to 1 year post KP | From pre-operation to 1 year post KP
  Weight for height (length) Z-score is calculated based on the gender, age, and weight reference standards for children in China. The difference in weight for height (length) Z-score between pre-operation and 1 year post KP is regarded as weight gain.
Liver parameters at post-operation month 6 | 6 months after KP
  Liver parameters: pediatric end-stage liver disease (PELD) score, liver stiffness measurement.
  PELD score = 0.480×ln (total bilirubin) + 1.857×ln (international normalized ratio)-0.687×ln (albumin) + 0.436 × age score + 0.667 × growth arrest] × 10. Age score:1 point for age < 24 months, 0 for age ≥ 24 months. Growth arrest: 1 point for more than 2 standard deviations below the average, otherwise 0.
  Liver stiffness measurement is measured by liver transient elastography.
Liver parameters at post-operation month 12 | 1 year after KP
  Liver parameters: pediatric end-stage liver disease (PELD) score, liver stiffness measurement.
  PELD score = 0.480×ln (total bilirubin) + 1.857×ln (international normalized ratio)-0.687×ln (albumin) + 0.436 × age score + 0.667 × growth arrest] × 10. Age score:1 point for age < 24 months, 0 for age ≥ 24 months. Growth arrest: 1 point for more than 2 standard deviations below the average, otherwise 0.
  Liver stiffness measurement is measured by liver transient elastography.
Changes in intestinal flora from post-operation week 2 to month 3 | From post-operation week 2 to month 3
  Fecal samples of 40 patients in each group are collected 2 weeks and 3 months after KP, and frozen at -80℃. 16s-rDNA sequencing is used to find out the changes in intestinal flora.
Changes in intestinal flora from post-operation week 2 to month 6 | From post-operation week 2 to month 6
  Fecal samples of 40 patients in each group are collected 2 weeks and 6 months after KP, and frozen at -80℃. 16s-rDNA sequencing is used to find out the changes in intestinal flora.

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Calinescu AM, Madadi-Sanjani O, Mack C, Schreiber RA, Superina R, Kelly D, Petersen C, Wildhaber BE. Cholangitis Definition and Treatment after Kasai Hepatoportoenterostomy for Biliary Atresia: A Delphi Process and International Expert Panel. J Clin Med. 2022 Jan 19;11(3):494. doi: 10.3390/jcm11030494. PMID 35159946
- [Background] Chen G, Liu J, Huang Y, Wu Y, Lu X, Dong R, Shen Z, Sun S, Jiang J, Zheng S. Preventive effect of prophylactic intravenous antibiotics against cholangitis in biliary atresia: a randomized controlled trial. Pediatr Surg Int. 2021 Aug;37(8):1089-1097. doi: 10.1007/s00383-021-04916-z. Epub 2021 May 19. PMID 34013444
- [Background] Decharun K, Leys CM, West KW, Finnell SM. Prophylactic Antibiotics for Prevention of Cholangitis in Patients With Biliary Atresia Status Post-Kasai Portoenterostomy: A Systematic Review. Clin Pediatr (Phila). 2016 Jan;55(1):66-72. doi: 10.1177/0009922815594760. Epub 2015 Jul 15. PMID 26183324
- [Background] Vangay P, Ward T, Gerber JS, Knights D. Antibiotics, pediatric dysbiosis, and disease. Cell Host Microbe. 2015 May 13;17(5):553-64. doi: 10.1016/j.chom.2015.04.006. PMID 25974298